CLINICAL TRIAL: NCT06584786
Title: Therapeutic Effects of Jing Si Herbal Tea for Chronic Obstructive Pulmonary Disease: A Comprehensive Investigation From Clinical to Basic Research
Brief Title: Therapeutic Effects of Jing Si Herbal Tea for COPD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-XD-132
Record Dates: First submitted 2024-04-02; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Airway Disease
Keywords: COPD; Jing Si herbal tea; damage-associated molecular patterns
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: In the COPDAE part, the control group received standard treatment including intravenous steroids, inhaled butanyl and ipratropium, and parenteral antibiotics for secondary infections. Placebo mimics of JSHT were administered to the control group. The JSHT group received standard COPDAE treatment plus JSHT (1 pack thrice daily) for one week. For patients with stable COPD, the control group received standard inhaled medications according to the GOLD guidelines. Placebo mimics of JSHT were administered to the control group. The JSHT group additionally received one pack of JSHT daily for three months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo group (1) (Placebo Comparator): Placebo group: participants with COPD AE is treated with placebo that mimic JSHT
  Interventions: Other: Placebo
- Placebo group (2) (Placebo Comparator): participants with stable COPD treated with placebo that mimic JSHT
  Interventions: Other: Placebo
- JSHT group of stable COPD (Experimental): participants with stable COPD treated with JSHT
  Interventions: Combination Product: Jing Si herbal tea (JSHT)
- JSHT group of COPDAE (Experimental): participants with COPD AE is treated with JSHT
  Interventions: Combination Product: Jing Si herbal tea (JSHT)

INTERVENTIONS:
Combination Product: Jing Si herbal tea (JSHT) — JSHT has been approved by the Ministry of Health and Welfare of Taiwan (registration number MOHW-PM-060635).
  Arms: JSHT group of COPDAE; JSHT group of stable COPD
Other: Placebo — Placebo of JSHT
  Other Names: Placebo of JSHT
  Arms: Placebo group (1); Placebo group (2)

SUMMARY:
Chronic obstructive pulmonary disease (COPD), a leading cause of global mortality, significantly impairs health-related quality of life (HRQL). COPD is characterized by airway inflammation and lung tissue damage. Jing Si herbal tea (JSHT) is known to have anti-inflammatory effects but has not been explored for treating COPD. This study investigated the potential of JSHT as an adjuvant therapy for COPD. This randomized controlled study focused on patients with COPD in the exacerbation and stable phases. The control group received the standard treatment, and the JSHT group received the standard treatment plus JSHT. Both groups underwent HRQL assessments, blood tests, and cellular studies involving five different groups to assess the effect of JSHT on damage-associated molecular patterns (DAMPs) and inflammatory markers.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common lung disease that impairs airflow and causes breathing difficulties. COPD is a major contributor to chronic health issues and mortality globally; it ranked as the third leading cause of death worldwide, resulting in 3.23 million fatalities in 2019. Individuals with COPD typically develop lung damage or airway obstruction. This condition is characterized by several common symptoms, including coughing, phlegm production, difficulty breathing, wheezing, and fatigue. The challenge in breathing frequently leads to reduced exercise endurance and diminished daily activity levels, which negatively affects health-related quality of life (HRQL). Despite following the optimal treatment provided by the Global Initiative for chronic obstructive lung disease (GOLD) guidelines, patients with COPD still experience significant disease effects. This underscores the need for continued research on potential therapies for COPD.

COPD is a gradually progressive airway disease. Harmful agents such as cigarettes and infection are the primary risk factor for COPD. The development of COPD involves airway inflammation and damage to the lung tissue. Persistent exposure to harmful agents damages lung epithelial cells, playing a crucial role in the pathogenesis of COPD. During this process, damage-associated molecular patterns (DAMPs) are released, triggering inflammatory pathways and the release of pro-inflammatory cytokines such as interleukin (IL)-1, IL-6, IL-8, and tumor necrosis factor (TNF)-α. These cytokines further activate inflammatory cells, such as macrophages and neutrophils, leading to further damage to lung tissues. These inflammatory mechanisms offer insights into potentially effective treatments.

Jing Si Herbal Tea (JSHT) is a herbal blend formulated to regulate the immune system and treat inflammatory respiratory conditions. A recent study showed that combining JSHT with standard treatment in patients with COVID-19 improved clinical C-reactive protein levels and alleviated infections more effectively than standard treatment alone. Additionally, using JSHT decreases the risk of intubation, critical conditions, and mortality. This suggests that JSHT may be a beneficial adjunct therapy for patients with COVID-19. However, the therapeutic effects of JSHT in COPD have not yet been studied.

Given that JSHT was designed for immune regulation and treatment of inflammatory diseases, investigators hypothesized that JSHT could be beneficial for patients with COPD. Therefore, investigators study the therapeutic effects and precise mechanisms of action of JSHT in COPD. This study provides a possible strategy for using JSHT as an adjuvant therapy for COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients willing to enter this study

Exclusion Criteria:

* not COPD patients, no willing to enter this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | Assess at baseline and three months of treatment
  The Taiwan Society of Pulmonary and Critical Care Medicine offers the Chinese version of the COPD Assessment Test (CAT) on the website (http://tspccm.org.tw). This test consists of eight items designed to evaluate COPD symptoms. These symptoms include cough, phlegm production, chest tightness, breathlessness, limitations in daily activities, confidence in leaving the house, sleep disturbances, and energy levels. Each symptom is rated on a scale from 0 to 5, culminating in a total CAT score ranging from 0 to 40. A higher score reflects more severe COPD symptoms. A score of 10 or higher is indicative of a significant symptom burden.
Modified Medical Research Council (mMRC) | Assess at baseline and three months of treatment
  The Modified Medical Research Council (mMRC) scale was used to evaluate dyspnea. This scale, comprising a 5-point grading system ranging from 0 to 4, measures dyspnea severity. A score of 0 indicates dyspnea only during intense exercise, while a sore of 4 represents breathlessness at rest.
Brief Symptom Rating Scale (BSRS-5) | Assess at baseline and three months of treatment
  The 5-item Brief Symptom Rating Scale (BSRS-5) was used to assess psychological distress. It consists of five items: feeling tense, being easily angered, feeling depressed, feeling inferior to others, difficulty with sleep, and suicidal thoughts. The scale is a 5-point scale ranging from 0 (not at all) to 4 (extremely), with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chou-Chin Lan, MD, Principal Investigator — Taichung Tzu Chi Hospital; Yao-Kuang Wu, MD, Study Director — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Xindan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The research is ongoing and not suitable for publication in order to protect intellectual property.

DOCUMENTS (3):
  • Study Protocol (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT06584786/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT06584786/SAP_001.pdf
  • Informed Consent Form (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT06584786/ICF_002.pdf